CLINICAL TRIAL: NCT00554398
Title: Impact of MK-0518 (Raltegravir) Intensification on HIV-1 Viral Latency in Patients With Previous Complete Viral Suppression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTEGRAL
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Raltegravir; MK-0518; Treatment intensification; HIV-1 latency; HIV eradication; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): MK-0518 400mg twice a day
  Interventions: Drug: MK-0518 400mg twice a day
- B (No Intervention): No intervention

INTERVENTIONS:
Drug: MK-0518 400mg twice a day — Raltegravir, MK-0518
  Other Names: Raltegravir
  Arms: A

SUMMARY:
An intensification with the HIV-1 integrase inhibitor Raltegravir (RAL) of a stable HAART regimen with persistent HIV-1 viral suppression could increase the slope of decay of the HIV-1 latent reservoir.

DETAILED DESCRIPTION:
While highly active antiretroviral therapy (HAART) reduces plasma HIV-1 levels to below the limits of detection with standard assays, replication-competent virus persist in a stable, latent reservoir in resting CD4+ T cells. So, there is a rapid resumption in plasma viremia when therapy is interrupted.

In addition to cellular reservoir, other pharmacologically privileged areas such as the central nervous system and the genital tract might act as additional sources of residual virus in patients with undetectable levels of plasma HIV-1 RNA. There is great current interest in strategies for depleting and eliminating this reservoir.

The antiviral potency of current regimens emerges as an important determinant of complete viral control. In certain patients, the latent reservoir decay can be hastened with treatment intensification.

An intensification with the HIV-1 integrase inhibitor Raltegravir (RAL) of a stable HAART regimen with persistent HIV-1 viral suppression could increase the slope of decay of the HIV-1 latent reservoir. This could provide further insight into this area, decrease the size of latent reservoir, and translate into clinical benefits for patients being simplified to maintenance monotherapy with RAL or in the HIV-1 rebound kinetics and slope after a programmed treatment interruption.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults (+18 years old).
2. Complete virological suppression (<50 copies/mL) for += 12 months, including at least 3 times during the last year.
3. Patients on HAART regimen including a PI or an NNRTI and at least two nucleotide inhibitors.
4. Voluntary written informed consent.

Exclusion Criteria:

1. Pregnancy, or fertile women willing to be pregnant.
2. Active substance abuse or major psychiatric disease.
3. Presence of drug-related mutations or any polymorphism or mutation associated to MK-0518 resistance prior to first HAART (only if genotype is available).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Quantification of integrated and unintegrated viral HIV-1 DNA in PBMCs | Basal, week 12, week 24 and week 48

SECONDARY OUTCOMES:
Quantification of residual HIV-1 (using an ultrasensitive RT-PCR assay with a lower limit of quantification of 5 copies/mL) | Basal, week 1, week 2, week 4, week 8, week 12, week 24, week 36 and week 48
Blips during the study (> 50 copies/mL, preceded and followed by determinations < 50 copies/mL in previous and posterior controls) | Basal, week 4, week 8, week 12, week 24, week 36 and week 48
Lymphocyte activation marker CD8+HLADR+CD38+ | Basal, week 2, week 4, week 12, week 24 and week 48.
Raltegravir plasma trough concentration. | Week 12, week 24 and week 48
Level of apoptosis in CD4 and CD8 T cells. | Week 48 and week 60

CONTACTS AND LOCATIONS:
Overall Officials: Martínez-Picado Javier, MD,PhD, Principal Investigator — Irsi Caixa -Hospital Germans Trias i Pujol; Paredes Roger, MD,PhD, Principal Investigator — Lluita contra la Sida Foundation; Clotet Bonaventura, MS,PhD, Principal Investigator — Lluita contra la Sida Foundation; Llibre Josep Mª, MD,PhD, Study Director — Lluita contra la SIDA Foundation
Locations (3):
- Spain (3):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clínic I Provinical de Barcelona, Barcelona

REFERENCES:
- [Derived] Llibre JM, Buzon MJ, Massanella M, Esteve A, Dahl V, Puertas MC, Domingo P, Gatell JM, Larrouse M, Gutierrez M, Palmer S, Stevenson M, Blanco J, Martinez-Picado J, Clotet B. Treatment intensification with raltegravir in subjects with sustained HIV-1 viraemia suppression: a randomized 48-week study. Antivir Ther. 2012;17(2):355-64. doi: 10.3851/IMP1917. Epub 2011 Sep 28. PMID 22290239